CLINICAL TRIAL: NCT04075630
Title: Observatory on Different Artificial Labour-induction Methods and Measuring Immediate Postpartum Maternal Satisfaction
Brief Title: Observatory on Artificial Labour-induction Methods and Measuring Immediate Postpartum Maternal Satisfaction
Acronym: SATISFACC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2018-03/BC-01
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Labor Induction
Keywords: childbirth; oxytocin; prostaglandin; cervical ripening balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Our hypothesis is that there is one sequence of labour-induction that leads to a better experience of childbirth than others. This is based on the following underlying theories :

* Maternal satisfaction depends on the number of labour-inducing sequences
* A longer labour-induction would be experienced less positively than a shorter one
* The experience is correlated with maternal outcomes ( vaginal / Caesarian delivery, spontaneous birth or instrument-assisted birth, maternal complications ) and neonatal outcomes (neonatal complications, secondary hospitalization).

DETAILED DESCRIPTION:
Artificial labour induction is a medical intervention used in the interest of the mother or unborn child, aimed at provoking birth by inducing uterine contractions artificially, leading to cervical effacement and dilation. The purpose is to end the pregnancy in the interest of the mother and/or foetus.

According to the latest results of the Perinatal Enquiry (2016), induced labour rates total around 22% of pregnancies (767.000 births in 2017) in all maternity clinics. For the university hospitals of Nimes and Montpellier, with Level 3 maternity units (thus requiring a higher rate of inductions), this represents 515 and 550 pregnancies respectively (2017 figures).

There are several methods of inducing labour: use of a cervical ripening balloon (a medical device with which the onset of labour is provoked mechanically), vaginal inserts containing prostaglandins or intravenous perfusion with oxytocin combined with water-breakage. These labour-induction methods may be used alone or in succession depending on the evaluation of the cervix using the Bishop score as a reference. Each method has its own benefits and risks.

There is variability between establishments in the protocols used for cervical ripening.

The Nimes and Montpellier centres both use the same methods, but with different sequences.

Studies are mainly devoted to evaluating each method individually in terms childbirth by vaginal delivery and duration of labour.

Maternal satisfaction, which is a rarely studied multifactorial evaluation, is correlated with women's psychological outcome. A bad experience during childbirth appears to increase the risk of post-partum (PP) psychological disorders.

Considering the current literature available, although there have been trials comparing two isolated labour-induction methods, like the study by Probaat (Jozwiak et al., 2013), which compared obstetrical and neonatal outcomes with the cervical ripening balloon and the prostaglandin insert, none of these studies investigated their impact on maternal satisfaction. Although there have been a few studies evaluating maternal satisfaction at childbirth, there have not been any evaluating satisfaction during artificial labour-induction in a pragmatic situation.

The aim of our study was therefore to evaluate the impact on semi-immediate maternal satisfaction under pragmatic, real-life conditions depending on the various possible induction scenarios (both in terms of the number of methods used, from 1 to 3, and the possible combinations when at least 2 or more methods were used ).

ELIGIBILITY:
Inclusion Criteria:

The patient has made no formal opposition to taking part in the study.

* The patient must be affiliated to/have the benefit of a health insurance scheme.
* The patient is at least 18 years old.
* The patient is capable of understanding the instructions required for answering questionnaires in French.

Concerning the targeted population:

* The patient has a medical indication for labour-induction.
* Term ≥ 37 weeks.
* The foetus is alive and viable, without any known lethal pathology

Exclusion Criteria:

The person is in a period of exclusion determined by a previous study.

* The person has been placed under judicial protection and is under guardianship or curatorship.
* It is impossible to give the person accurate information.

Non-inclusion criteria concern associated illnesses or interfering conditions:

* The patient does not have the possibility to answer the questionnaire at 1 month
* Contra-indication for labour-induction or vaginal delivery
* Foetal presentation other than cephalic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women at the end of pregnancy
Study Population: Women 18+ admitted to gynecology-obstetric depts. of Montpellier & Nîmes University Hospitals for artificial labor-induced childbirth. Sociodemographic and medical variables will be noted: patient's knowledge of labor-induction, labor in childbirth, age, weight, height (BMI), no. of previous pregnancies, childbirths, miscarriages, abortions, medically-motivated induced terminations, medical antecedents (comorbidities), important surgery (esp. uterine), ongoing treatment, tobacco/alcohol/cannabis intake, Down's syndrome screening, pregnancy particularities (medically-assisted procreation), antenatal diagnosis, no. of hospital consultations, gestational age at admission, information received, other newborn data (term, weight, size, cranial perimeter at birth), reason for induction.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction | 2 hours after giving birth
  Overall patient satisfaction evaluated via a 4-point Likert scale (1= not satisfied, 2 = moderately satisfied, 3 = satisfied, 4 = very satisfied) on a touchscreen.

SECONDARY OUTCOMES:
Patient satisfaction evaluated via the W-DEQ questionnaire | 2 hours after giving birth
  The Wijma Delivery Experience Questionnaire (W-DEQ) is a Scandinavian questionnaire (designed by Wijma et al. in 1998) translated into French. It evaluates the patient's true experience of childbirth compared with her expectations. It has 33 items based on recurring fears of pregnant women, divided into several catégories (fear, negative feelings, lack of confidence, behaviour etc…).
Post-partum QEVA satisfaction questionnaire | 1-2 months after giving birth
  The pluridimensional Questionnaire d'Evaluation du Vécu de l'Accouchement (QEVA) known in English as the QACE (Questionnaire for Assessing the Childbirth Experience is used to evaluate the patient's experience of childbirth. It contains 25 items, each with a 4-point Likert scale, divided into the following categories: relationship with healthcare teams, emotions (positive and negative), first moments with the newborn baby, situation one month after childbirth. An e-mail is sent to the patient 1 month after giving birth, asking her to complete the QEVA by logging onto a dedicated platform.
Different methods of labour-induction used | 6 months after giving birth
  Data collection from medical files on the methods of labour-induction used (alone or successively), duration of use and intermediate Bishop scores. This a pre-labor scoring system reflecting cervical modification ranges from 0 to 3 (0= cervix closed and 3 = dilated to more than 5 cm) assists in predicting whether labour-induction will be required and the likelihood of spontaneous preterm delivery.
Spontaneous vaginal deliveries | 48 hours maximum
  Rate of spontaneous vaginal deliveries,
Rate of instrument-assisted vaginal deliveries | 48 hours maximum
  Rate of instrument-assisted vaginal deliveries.
Reason for instrument-assisted vaginal deliveries | 48 hours maximum
  Reason for instrument-assisted vaginal deliveries (non progression of fœtal presentation, fœtal distress, maternal complications).
Type of instrument-assisted vaginal deliveries | 48 hours maximum
  Type of instrumental extraction used for the delivery
  .
Rate of Caesarian births | 48 hours maximum
  Rate of Caesarian births and reason (no cervical dilatation at the first stage of labour : dilatation 0 to 10cm, absence of fœtal descent at stage 2 of labour, fœtal cause, maternal cause).
Reason for Caesarian births | 48 hours maximum
  Reason for Caesarian birth (no cervical dilatation at the first stage of labour : dilatation 0 to 10cm, absence of fœtal descent at stage 2 of labour, fœtal cause, maternal cause).
Time from start of labour-induction to start of labour | 48 hours maximum
  Time between the start of labour-induction and the onset of labour will be measured
Time from labour-induction to birth (Caesarian births excluded), | 48 hours maximum
  Time from labour-induction to vaginal delivery
Vaginal deliveries at H12 | 12 hours from start of induction
  Rate of vaginal deliveries at 12 hours from start of labour-induction
Vaginal deliveries at H24 | 24 hours from start of induction
  Rate of vaginal deliveries at 24 hours from start of labour-induction
Vaginal deliveries at H48 | 48 hours from start of induction
  Rate of vaginal deliveries at 48 hours from start of labour-induction
Labour-induction failures | 12 - 18 hours
  Rate of labour-induction failures giving rise to a Caesarian due to the duration of the latency phase (0-6cm) ≥24h with oxytocine administered for at least 12-18h after artificial water-breakage.
Propess | up to 48 hours before birth
  Rate of secondary or tertiary use of Propess (vaginal prostaglandine inserts)
Balloon/Foley bulb | 48 hours maximum
  Rate of secondary or tertiary use of the cervical ripening balloon (Foley bulb)
Oxytocine | 48 hours maximum
  Rate of secondary or tertiary use of intravenous Oxytocine
Epidurals | 48 hours maximum
  Rate of epidural anesthaesia during labour
Bishop score evolution: Propess | Until birth (48 hours maximum)
  The Bishop score,developed by Professor Emeritus of Obstetrics and Gynecology Dr. Edward Bishop, is also known as cervix score. It is a pre-labor scoring system to assist in predicting whether induction of labor will be required. It is based on 5 points : Cervical dilation in centimeters, cervical effacement as a percentage,cervical consistency by provider assessment/judgement, cervical position, fetal station (the position of the fetal head in relation to the pelvic bones).The Bishop score grades patients who would be most likely to achieve a successful induction. The duration of labor is inversely correlated with the Bishop score; a score that exceeds 8 describes the patient most likely to achieve a successful vaginal birth. Bishop scores of less than 6 usually require a cervical ripening method (pharmacologic or physical, such as a Foley bulb).
Bishop score evolution: Balloon/Foley bulb | Until birth (48 hours maximum)
  The Bishop score,developed by Professor Emeritus of Obstetrics and Gynecology Dr. Edward Bishop, is also known as cervix score. It is a pre-labor scoring system to assist in predicting whether induction of labor will be required. It is based on 5 points : Cervical dilation in centimeters, cervical effacement as a percentage,cervical consistency by provider assessment/judgement, cervical position, fetal station (the position of the fetal head in relation to the pelvic bones).The Bishop score grades patients who would be most likely to achieve a successful induction. The duration of labor is inversely correlated with the Bishop score; a score that exceeds 8 describes the patient most likely to achieve a successful vaginal birth. Bishop scores of less than 6 usually require a cervical ripening method (pharmacologic or physical, such as a Foley bulb).
Bishop score evolution: Ocytocine | Until birth (48 hours maximum)
  The Bishop score,developed by Professor Emeritus of Obstetrics and Gynecology Dr. Edward Bishop, is also known as cervix score. It is a pre-labor scoring system to assist in predicting whether induction of labor will be required. It is based on 5 points : Cervical dilation in centimeters, cervical effacement as a percentage,cervical consistency by provider assessment/judgement, cervical position, fetal station (the position of the fetal head in relation to the pelvic bones).The Bishop score grades patients who would be most likely to achieve a successful induction. The duration of labor is inversely correlated with the Bishop score; a score that exceeds 8 describes the patient most likely to achieve a successful vaginal birth. Bishop scores of less than 6 usually require a cervical ripening method (pharmacologic or physical, such as a Foley bulb).
Maternal morbidity | 6 months after giving birth
  Rate of uterine hyperstimulation(> 6 contractions in 10 minutes on 2 occasions) with or without an effect on the foetus
Maternal morbidity | 48 hours maximum
  Rate of uterine hypertonia (contraction > 2 minutes with slowing down of fœtal heartbeat)
Maternal morbidity: moderate haemorrhage | 48 hours maximum
  Rate of post partum haemorrage ≥ 500ml, rate of severe post-partum haemorrhage ≥1000ml, rate of transfusion, number of packs of red blood cells transfused
Maternal morbidity: severe haemorrage | 48 hours maximum
  rate of severe post-partum haemorrage ≥1000ml rate of transfusion, number of packs of red blood cells transfused
Maternal morbidity: transfusion rate | 48 hours maximum
  Rate of transfusions
Maternal morbidity: amount of blood transfused | 48 hours maximum
  This is measured in terms of the number of packs of red blood cells transfused
Maternal morbidity: rupture | 48 hours maximum
  Rate of uterine rupture
Maternal morbidity: Chorioamniotitis | 48 hours maximum
  Chorioamniotitis (temperature > 38°C with fœtal tachycardia > 160 beats / minute)
Maternal morbidity: infection | 1 week after giving birth
  Rate of post-partum infection (temperature > 38°C with antibiotherapy, urinary infection, bacteriologically-proven endometritis at 1 week post-partum)
Neonatal morbidity:asphyxia | 5 minutes after giving birth
  Rate of neonatal asphyxia (umbilical cord arterial pH ≤ 7.05, and/or APGAR at 5 minutes < 7). The Apgar score is a means of evaluating the vitality of a newborn based on the simple observation at the time of birth. The value is a prognostic for neonatal mortality. It was developed in 1952 by the American doctor, Virginia Apgar.
Neonatal morbidity: neonatal hospitalisation | up to 48 hours after giving birth
  Rate of neonatal pediatric hospitalisations
Neonatal morbidity: infection | up to 48 hours after giving birth
  Bacteriologically-proven infection rate
Maternal tolerance: bleeding | up to 48 hours after giving birth
  Metrorrhagia due to vaginal insert (dinoprostone) or cervical ripening balloon placement
Maternal tolerance: pain due to overinflation of the balloon (Foley bulb) | up to 48 hours after giving birth
  Pain related to balloon inflation requiring secondary partial deflation, reorded with a VAS. The visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity
Maternal tolerance: pain on 1st induction sequence | up to 48 hours before birth
  Pain level recorded with a VAS before the 1st induction sequence. The visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity
Maternal tolerance: pain after childbirth | 2 hours after giving birth
  Pain level recorded with a VAS at H2 of childbirth.
Maternal tolerance: pain during childbirth | labour time
  Pain level at various times of labour-induction recorded with a VASThe visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity
Maternal tolerance: pain due to insert or balloon (Foley bulb) | up to 48 hours before birth
  Pain level recorded with a VAS before vaginal insert or balloon placement. The visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity
Maternal tolerance: pain due to insert or balloon (Foley bulb) at H2 | 2 hours after device placement
  Pain level recorded with a VAS 2 hours after vaginal insert or balloon placement. The visual analog scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: vincent letouzey, M., Principal Investigator — CHU de Nîmes Service de Gynécologie Obstétrique
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire, Nîmes, Gard
  - CHU Arnaud de Villeneuve Service de Gynécologie Obstétrique, Montpellier, Hérault